CLINICAL TRIAL: NCT05769114
Title: Outcome of Surgical Versus Primary Non-Surgical Treatment of Traumatic Thoracolumbar Spine Burst Fracture in Patients Without Neurological Symptoms: A Randomized Controlled Clinical Trial
Brief Title: Surgical Versus Non-Surgical Treatment of Thoracolumbar Burst Fracture
Acronym: A34RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00662
Record Dates: First submitted 2023-02-08; First posted 2023-03-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: SPINAL Fracture; Burst Fracture; Spinal Instability of Thoracolumbar Region
Keywords: Traumatic Thoracolumbar Spine Burst Fracture
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgical treatment (Active Comparator): The surgeon will perform a minimally invasive (percutaneous) posterior stabilization of the injured spinal segments. Transpedicular screws will be inserted into the vertebral body superior and inferior to the fractured vertebra under fluoroscopic control. In a second stage procedure a lumbo- or thoracotomy (depending on the fracture level below or above the diaphragm) is performed to remove the fractured part of the vertebral body (hemicorporectomy) including the intervertebral disc segments. The resulting void is replaced by an (expandable) spacer/cage.
  Interventions: Procedure: Surgical stabilization
- Non-surgical treatment (No Intervention): The patients will receive an external bracing (3-point hyperextension brace) for six weeks, which must be always worn except when lying flat in bed. The brace is adjusted by an experienced orthopedist. A physiotherapist will instruct the patient to accomplish daily activities with the restriction he or she will have by wearing the brace.
- Observational arm (Other): Patients who do not agree to randomization will be given the option to participate in the observational arm of the study. Their treatment will be surgical fixation with an anterior-posterior stabilization (as per our current internal hospital standard).
  Interventions: Procedure: Surgical stabilization

INTERVENTIONS:
Procedure: Surgical stabilization — Anterior-posterior stabilization (360°) with pedicle screws and an expandable cage
  Other Names: 360°-Stabilization
  Arms: Observational arm; Surgical treatment

SUMMARY:
Treatment for acute traumatic thoracolumbar burst fractures differs significantly across the world in patients without neurological impairments and without damage to the posterior column of the spine. This randomized controlled, non-inferiority clinical trial's goal is to evaluate the effectiveness of surgery versus initial non-surgical treatment for patients with traumatic thoracolumbar spine burst fractures who don't have any neurological symptoms.

The study's precise objectives are to:

1. evaluate the clinical outcome (Oswestry Disability Index)
2. evaluate the radiography result (restoration and maintenance of spinal alignment)
3. determine the prevalence of complications

at least 24 months of follow-up of neurologically unaffected patients with acute traumatic burst fractures. Both groups will get the same therapy using standardized methods: The surgical group's entire patient population will get combined anterior-posterior (360°) spinal fusion therapy. Three-point hyperextension orthoses will be used to treat all patients in the non-surgical group for six weeks following the injury.

DETAILED DESCRIPTION:
The research is a single-center, nationwide, randomized controlled trial. Over a two-year period, 52 patients with a thoracolumbar burst fracture will enroll in the study. They will be assigned randomly (1:1) to either non-surgical treatment with a brace or surgery with anterior-posterior fixation. A prospective data collection will be asked of subjects who decline randomization (observational arm). The subjects will be evaluated clinically, radiologically, and based on patient-reported outcomes over the course of two years. Both patient files and questionnaires will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years at inclusion
* Acute traumatic burst fracture of the thoracolumbar spine (10th thoracic to 3rd lumbar vertebral body)
* Informed consent for study participation

Exclusion Criteria:

* Injury of the posterior tension band/posterior column of the thoracolumbar spine
* Any neurological deficit (American Spinal Injury Association Impairment Scale [AISA] Grade A-D)
* Pathological vertebral body fractures (diagnosed by MRI and CT scan), which, in the opinion of the research/investigative team, would compromise (or interfere with) patients' ability to participate in the study
* Concomitant spinal fractures at any other level of the spine outside the T10-L3 level, which, in the opinion of the research/investigative team, would compromise (or interfere with) patients' ability to participate in the study
* Multiple trauma or Injury Severity Score (ISS) > 16 or additional injuries according to the investigator may, which, in the opinion of the research/investigative team, would compromise (or interfere with) patients' ability to participate in the study (impairment of early ambulation)
* Any known previous spinal surgery in the thoracolumbar spine, which, in the opinion of the research/investigative team, would compromise (or interfere with) patients' ability to participate in the study
* Any severe, progressive, or uncontrolled medical or psychiatric condition, or other factors at randomization that in the judgment of the investigator prevents the patient from participating in the study
* Known history of substance abuse (i.e., recreational drugs, alcohol) that would preclude reliable assessment in the opinion of the investigator
* Pregnancy or women planning to conceive within the study period. All women included in this study must have a negative blood pregnancy test (human chorionic gonadotrophin (hCG) blood level at visit 1. If pregnancy occurs during the study period, the patients drop out of the study
* Inability to follow the procedures of the study, e.g., due to inability to understand German, French or English, which, according to the investigator, may jeopardize the patient in case of participation in the study or prevents the patient from participating in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
The clinical outcome as assessed by the Oswestry Disability Index (ODI) 104 weeks post-surgery or non-surgical treatment initiation | 2 years after fracture
  ODI is a patient-reported outcome measure for spinal disorders. It consists of 10 questions related to back specific disabilities such as pain, personal care, walking and sitting ability, lifting capacity and social life.

SECONDARY OUTCOMES:
Radiological outcome: Mono- (A3-fractures)/Bisegmental (A4-fractures) kyphosis angle | Pre-Treatment to 2 years after the fracture
  Bi-/segmental kyphosis (Gardner/Cobb angle) assessed by long-standing x-rays of the entire spine
Radiological outcome: Spinal fusion and fracture consolidation | 26 weeks after fracture
  Spinal fusion in the surgical group and fracture consolidation in the non-surgical group assessed by CT-scan
Radiological outcome: Segment mobility | 52 weeks after fracture
  Segment mobility assessed by functional lateral views at 52 weeks and compared between treatment groups
Radiological outcome: Degeneration of the intervertebral disc over time | Pre-Treatment, 52 weeks after the fracture
  Degeneration of the intervertebral disc (Pfirrmann grade)
Radiological outcome: Progression of spinal canal stenosis | From the time of fracture, 26 weeks and 52 weeks
  Assessed on CT-scan and MRI
Non-surgical treatment failure rate | From the time of fracture to 2 years after the fracture
  Proportion/frequency of patients in the non-surgery group that received surgery later, if there is a clinical indication (spinal instability measured by a kyphosis > 30 degrees on x-ray, intolerable pain, delayed onset of neurological symptoms) or if the patient is not satisfied after treatment
Complication rate and severity and additional surgeries | 6, 12, 26, 52, and 104 weeks
  Rate and severity according to the Spine Adverse Events Severity System (SAVES) and surgical complications between treatment groups
Changes in patient-related outcome measurements: AOSpine Patient Reported Outcome Spine Trauma (PROST) | From the time of fracture to 2 years after the fracture
  Changes between groups and from baseline to follow-up 104 weeks and compared between treatment groups
Changes in patient-related outcome measurements: EQ5D-3L | Pre-Treatment to 2 years after the fracture
  Changes between groups and from baseline to follow-up 104 weeks and compared between treatment groups
Changes in patient-related outcome measurements: Pain visual analogue scale (VAS) | Pre-Treatment to 2 years after the fracture
  Changes between groups and from baseline to follow-up 104 weeks and compared between treatment groups
Indirect costs | 6, 12, 26, 52, and 104 weeks
  Assessed by indirect cost questionnaire and compared between treatment groups
Treatment data: Length of hospitalization (days) | Pre-Treatment to discharge from hospital
  Inhospital data records, comparison between treatment groups
Treatment data: blood loss during surgery (ml) | during surgery
  Inhospital data records
Treatment data: duration of surgery (hh: mm) | during surgery
  Inhospital data records
Time to return to work/sports | 6, 12, 26, 52, and 104 weeks
  Documented at each clinical follow-up as internal clinic standard of care, comparison between treatment groups
Radiological outcome: Sagittal and coronal alignment | 6, 12, 26, 52, and 104 weeks
  Assessed by long-standing x-rays of the entire spine, comparison between treatment groups
Opioid use | Pre-Treatment, 6, 12, 26, 52, and 104 weeks
  Use of oral intake of opioids, comparison between treatment groups and changes from baseline to 104 weeks

OTHER OUTCOMES:
Radiological outcome: Fracture comminution | Pre-Treatment
  Fracture comminution of the vertebral body
Radiological outcome: Classification of traumatic disc injury | Pre-treatment
  Sanders Classification

CONTACTS AND LOCATIONS:
Overall Officials: Christoph E Albers, PD Dr., Principal Investigator — Inselspital Bern, Department of Orthopaedic Surgery and Traumatology; Sonja Häckel, Dr., Study Director — Inselspital Bern, Department of Orthopaedic Surgery and Traumatology
Locations (2):
- Switzerland (2):
  - Inselspital, Bern
  - Ostschweizer Wirbelsaeulenzentrum Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No
No process has been defined yet how the sharing of the data should proceed

REFERENCES:
- [Background] Gnanenthiran SR, Adie S, Harris IA. Nonoperative versus operative treatment for thoracolumbar burst fractures without neurologic deficit: a meta-analysis. Clin Orthop Relat Res. 2012 Feb;470(2):567-77. doi: 10.1007/s11999-011-2157-7. Epub 2011 Nov 5. PMID 22057820
- [Background] Vaccaro AR, Oner C, Kepler CK, Dvorak M, Schnake K, Bellabarba C, Reinhold M, Aarabi B, Kandziora F, Chapman J, Shanmuganathan R, Fehlings M, Vialle L; AOSpine Spinal Cord Injury & Trauma Knowledge Forum. AOSpine thoracolumbar spine injury classification system: fracture description, neurological status, and key modifiers. Spine (Phila Pa 1976). 2013 Nov 1;38(23):2028-37. doi: 10.1097/BRS.0b013e3182a8a381. PMID 23970107
- [Background] Oner FC, Wood KB, Smith JS, Shaffrey CI. Therapeutic decision making in thoracolumbar spine trauma. Spine (Phila Pa 1976). 2010 Oct 1;35(21 Suppl):S235-44. doi: 10.1097/BRS.0b013e3181f32734. PMID 20881467
- [Background] Spiegl UJ, Fischer K, Schmidt J, Schnoor J, Delank S, Josten C, Schulte T, Heyde CE. The Conservative Treatment of Traumatic Thoracolumbar Vertebral Fractures. Dtsch Arztebl Int. 2018 Oct 19;115(42):697-704. doi: 10.3238/arztebl.2018.0697. PMID 30479250